CLINICAL TRIAL: NCT00435240
Title: Paleolithic Diet in the Treatment of Diabetes Type 2 in Primary Health Care
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lund University Hospital (Other)
Responsible Party: Dr Tommy Jönsson, Department of Clinical Sciences, Medical Faculty, Lund University Hospital, Sweden
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H4 726/2004
Record Dates: First submitted 2007-02-13; First posted 2007-02-14 (Estimated); Last update posted 2008-05-15 (Estimated); Status verified 2008-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Diet, Paleolithic

INTERVENTIONS:
Behavioral: Paleolithic diet

SUMMARY:
There is uncertainty about the optimal diet in the prevention and treatment of diabetes type 2. Earlier studies have generally focused on intakes of fat, protein, carbohydrate, fiber, fruit and vegetables. This study is based on another approach which compares foods that were available during human evolution with more recently introduced ones. The basic tenet from evolutionary biology is that if human physiology is less adapted to a relatively recently introduced diet based on agriculture, this could cause disturbances to human physiology and ultimately lead to diseases. Epidemiological studies indicates that diabetes mellitus type 2 is absent or near absent in populations eating a Palaeolithic ("Old Stone Age") diet which is free from food items produced in agriculture or the food industry. Our study hypothesis is that a Palaeolithic diet is better than the standard diabetes diet recommended today in treating diabetes type 2.

Fifteen patients with diabetes type 2 have been randomized to

1. a Palaeolithic diet based on lean meat, fish, fruit, vegetables, root vegetables, eggs, and nuts
2. a standard diabetes diet as recommended by national health authorities.

The patients eat the diet they have been randomized to for three months and then switches to the other diet for another three months. The study is conducted in Primary Health Care stations.

ELIGIBILITY:
Inclusion Criteria:

* Adults with capacity to perform study
* Diabetes Mellitus Type 2
* C-peptide > 0
* HbA1C >5.5
* Unchanged diabetes treatment during last 3 months
* Weight and HbA1C varied less than 5% during last 3 months
* No acute heart disease during last 6 months
* Unchanged treatment with betablocker last 6 months
* Unchanged treatment with thyroid hormone substitution last 6 months

Exclusion Criteria:

* Treatment with insulin
* Chronic treatment with steroids (not inhaled)
* Treatment with Waran (anticoagulant cumarin type)
* Creatinin > 130 micromol/L
* Elevated liver enzymes (ALAT,ASAT,ALP or GT > 4 X upper reference value)
* Acute heart disease
* Changed treatment with betablocker or thyroid hormone substitution

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2005-01; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
area under the curve for glucose (AUC Glucose0-120) at the oral glucose tolerance test at baseline, 3 months and 6 months
area under the curve for insulin (AUC Insulin0-120) at the oral glucose tolerance test at baseline, 3 months and 6 months
HbA1C at baseline, 3 months and 6 months
weight at baseline, 3 months and 6 months
waist circumference at baseline, 3 months and 6 months

SECONDARY OUTCOMES:
satiation measured on visual semi-analogous scale at food intake during 4 days av 6 weeks and 12 weeks
leptin at baseline, 3 months and 6 months
fasting plasma glucose at baseline, 3 months and 6 months
fasting plasma insulin at baseline, 3 months and 6 months
Systolic and diastolic blod pressure at baseline, 3 months and 6 months
Blood lipids at baseline, 3 months and 6 months
C-reactive protein at baseline, 3 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Tommy Jönsson, MD, Principal Investigator — Department of Clinical Sciences, Lund University, Lund Sweden
Locations (1):
- Lund University Hospital, Lund, Skåne County, Sweden

REFERENCES:
- [Background] Jonsson T, Ahren B, Pacini G, Sundler F, Wierup N, Steen S, Sjoberg T, Ugander M, Frostegard J, Goransson L, Lindeberg S. A Paleolithic diet confers higher insulin sensitivity, lower C-reactive protein and lower blood pressure than a cereal-based diet in domestic pigs. Nutr Metab (Lond). 2006 Nov 2;3:39. doi: 10.1186/1743-7075-3-39. PMID 17081292
- [Background] Jonsson T, Olsson S, Ahren B, Bog-Hansen TC, Dole A, Lindeberg S. Agrarian diet and diseases of affluence--do evolutionary novel dietary lectins cause leptin resistance? BMC Endocr Disord. 2005 Dec 10;5:10. doi: 10.1186/1472-6823-5-10. PMID 16336696
- [Background] Cordain L, Eaton SB, Sebastian A, Mann N, Lindeberg S, Watkins BA, O'Keefe JH, Brand-Miller J. Origins and evolution of the Western diet: health implications for the 21st century. Am J Clin Nutr. 2005 Feb;81(2):341-54. doi: 10.1093/ajcn.81.2.341. PMID 15699220
- [Derived] Fontes-Villalba M, Granfeldt Y, Sundquist K, Memon AA, Hedelius A, Carrera-Bastos P, Jonsson T. Effects of a Paleolithic diet compared to a diabetes diet on leptin binding inhibition in secondary analysis of a randomised cross-over study. BMC Endocr Disord. 2024 Sep 4;24(1):176. doi: 10.1186/s12902-024-01715-0. PMID 39232748
- [Derived] Fontes-Villalba M, Lindeberg S, Granfeldt Y, Knop FK, Memon AA, Carrera-Bastos P, Picazo O, Chanrai M, Sunquist J, Sundquist K, Jonsson T. Palaeolithic diet decreases fasting plasma leptin concentrations more than a diabetes diet in patients with type 2 diabetes: a randomised cross-over trial. Cardiovasc Diabetol. 2016 May 23;15:80. doi: 10.1186/s12933-016-0398-1. PMID 27216013
- [Derived] Jonsson T, Granfeldt Y, Ahren B, Branell UC, Palsson G, Hansson A, Soderstrom M, Lindeberg S. Beneficial effects of a Paleolithic diet on cardiovascular risk factors in type 2 diabetes: a randomized cross-over pilot study. Cardiovasc Diabetol. 2009 Jul 16;8:35. doi: 10.1186/1475-2840-8-35. PMID 19604407